CLINICAL TRIAL: NCT02471092
Title: The Effect of Milk Proteins on Satiety, Food Intake and Metabolic Control (Glycemia) in Early Adulthood
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Guelph (Other)
Collaborators: University of Toronto (Other); Laval University (Other)
Responsible Party: Principal Investigator, Amanda Wright, Ph.D., Associate Professor, University of Guelph
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 14JN004
Record Dates: First submitted 2015-05-26; First posted 2015-06-15 (Estimated); Last update posted 2016-10-25 (Estimated); Status verified 2016-10

CONDITIONS: Hyperglycemia; Lack of Satiety
Keywords: satiety; glycemia; milk protein
MeSH Terms: conditions — Hyperglycemia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (5):
- Water Control (Placebo Comparator): Skim milk products. Water and permeate control; 250mL serving.
  Interventions: Other: Skim milk products
- Skim Milk (Active Comparator): Skim milk products. Skim milk (regular 80:20 protein ratio); 250mL serving.
  Interventions: Other: Skim milk products
- High Protein Milk (Experimental): Skim milk products. High protein milk (regular 80:20 protein ratio); 250mL serving.
  Interventions: Other: Skim milk products
- High Protein Milk (Modified Ratio) (Experimental): Skim milk products. High protein milk with modified protein ratio (40:60 ratio); 250 mL serving.
  Interventions: Other: Skim milk products
- Skim Milk (Modified Ratio) (Experimental): Skim milk products. Skim milk with modified protein ratio (40:60 ratio); 250 mL serving.
  Interventions: Other: Skim milk products

INTERVENTIONS:
Other: Skim milk products — Milk treatments will be served with 58g of breakfast cereal.

SUMMARY:
The purpose of this study is to develop and test modified milk protein products to determine the effects of amino acids on food intake, satiety, insulin secretion and glucose control by insulin-independent action in healthy adults.

DETAILED DESCRIPTION:
1. A total of 33 males and females will participate in the study. Capillary blood samples will be collected from all participants to measure plasma glucose over a 3.5 hour postprandial study.
2. Intravenous blood samples will be collected from a subset of 12 (6 males and 6 females) participants for determination of insulin, satiety hormones, acetaminophen (gastric emptying rates), and determination of amino acid profiles.

ELIGIBILITY:
Inclusion Criteria:

* BMI 20 - 24.9 kg/m2
* Healthy as determined by screening questionnaire
* Male or Female
* Non-smoking
* Normal fasting plasma glucose (<5.5 mmol/L), but not below 3.3 mmol/L.
* Prior use of acetaminophen

Exclusion Criteria:

* Gastrointestinal conditions or illness (including, but not limited to, lactose intolerance, Celiac, Crohn's, Ulcerative Colitis (UC), Irritable Bowel Disorder (IBD)
* Weight loss or weight gain of more than 5 kg during the previous 2 months
* Taking medication or protein supplements (excluding oral contraceptive, multivitamins and folic acid)
* Serious medical condition (ie. Renal, liver)
* Lack of appetite or skipping breakfast
* Restrained eaters as defined as having a Three Factor Eating Questionnaire-Cognitive Restraint >16
* Smoking
* Reported intolerance to milk or very low consumption (< 2 servings per week) as assessed by in-person screening. Or not liking of the research foods.
* Food allergies or intolerances as well as anaphylactic or life-threatening allergies - food or otherwise
* Diabetes or other metabolic diseases that could interfere with study outcomes
* Acetaminophen, codeine or opioid allergy
* Pregnant or Breast Feeding
* Typical alcohol consumption of not more than 4 drinks per sitting

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2014-11; Primary Completion 2015-10 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Postprandial Glycemia, as measured by capillary blood glucose (mmol/L) | 0-200 minutes

SECONDARY OUTCOMES:
Postprandial Satiety, as measured by paper 100-mm visual analogue scale (mm) | 0-200 minutes
Food Intake at ad libitum lunch meal, as measured by weighed pizza consumption (g) | at 120 minutes

OTHER OUTCOMES:
Hormone and Amino Acid Analysis, as measured by biochemical assay (pmol/L and nmol/mL) | 0-200 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Amanda J Wright, Ph.D., Principal Investigator — University of Guelph
Locations (1):
- University of Guelph- Human Nutraceutical Research Unit, Guelph, Ontario, Canada

REFERENCES:
- [Derived] Kung B, Turgeon SL, Vien S, Kubant R, El Khoury D, Wright AJ, Goff HD, Anderson GH. Role of Amino Acids in Blood Glucose Changes in Young Adults Consuming Cereal with Milks Varying in Casein and Whey Concentrations and Their Ratio. J Nutr. 2020 Dec 10;150(12):3103-3113. doi: 10.1093/jn/nxaa275. PMID 33024990